CLINICAL TRIAL: NCT05869162
Title: A Phase II, Open-Label, Single-Arm, Multicenter Study of Efficacy and Safety of SY-3505 in Patients With ALK-Positive Advanced Non-Small Cell Lung Cancer Who Have Progressed On or Are Intolerant to Second-Generation ALK TKI
Brief Title: Phase II Study of SY-3505 in Patients With ALK-positive NSCLC Who Have Failed Prior Second-Generation ALK TKI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shouyao Holdings (Beijing) Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-3505-II-01
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-05

CONDITIONS: Non-small-cell Lung Carcinoma
Keywords: SY-3505; Anaplastic lymphoma kinase; Non-small cell lung carcinoma; Third-generation ALK tyrosine kinase inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SY-3505-Phase II (Experimental): SY-3505 single agent, 600 mg oral capsules, QD, continuously
  Interventions: Drug: SY-3505

INTERVENTIONS:
Drug: SY-3505 — A Third-generation ALK TKI
  Other Names: CT-3505

SUMMARY:
This is an open-label, single-arm, multicenter, phase II study to evaluate the efficacy and safety of SY-3505 capsule in patients with locally advanced or metastatic NSCLC who have progressed on or are intolerant to second-generation ALK tyrosine kinase inhibitor (TKI).

DETAILED DESCRIPTION:
SY-3505 is a potent, brain-penetrant, third-generation ALK tyrosine kinase inhibitor (TKI) with preclinical activity against both wild-type and most known resistance mutations of ALK occurring in first-generation and second-generation ALK TKI-resistant patients.

In this phase 2 study, patients with locally advanced or metastatic NSCLC who have progressed on or are intolerant to second-generation ALK TKI will be treated with SY-3505 capsules at 600 mg once daily (QD) orally until disease progression, refusal or unacceptable toxicity. Cycles of treatment are every 21 days with continuous dosing of SY-3505. During the study, patients will be followed-up for safety and efficacy evaluation at study protocol defined time points.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible to participate in this study:

1. Age ≥ 18 years at the time of signing the informed consent form (ICF).
2. Histologically or cytologically confirmed locally advanced (tumor lesion could not be radically cued by surgery or radiation as asessed by the investigators) or metastatic NSCLC.
3. Prior treated with at least one second-generation ALK TKI (including unmarketed investigational drugs) and imaging evidence of disease progression (PD) or intolerance to prior treatment toxicity.
4. Agree to provide fresh tumor tissue samples to test positive for ALK fusion (ALK-positive) by the central laboratory:

   1. If the patient is indeed unable to provide fresh tumor tissue samples (e.g., repuncture has been assessed by the investigator as having a higher clinical risk) and cannot provide archived tissue samples within 2 years prior to initial administration, but can provide ALK-positive testing reports within 2 years prior to the first administration (detection methods include FISH, RT-PCR, IHC [Ventana method] or NGS, etc.), inclusion or not of the patient will be discussed and decided by the investigator and the sponsor;
   2. If the patient is indeed unable to provide either fresh tumor tissue samples (e.g., repuncture has been assessed by the investigator as having a higher clinical risk) or ALK-positive testing reports within 2 years prior to the first administration, but can provide archived tissue samples within 2 years prior to the first administration and confirmed as ALK-positive by the central laboratory, inclusion or not of the patient will be discussed and decided by the investigator and the sponsor.
5. Must have at least one extracranial target lesion that meets the RECIST 1.1 criteria; For a lesion that has previously received radiotherapy, it can be assessed as a target lesion only when it shows definite progression after radiotherapy.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
7. Estimated Life expectancy ≥ 3 months.
8. Prior antitumor treatment-related AE had recovered to ≤ Grade 1 as defined by NCI-CTCAE v 5.0 prior to initial administration (except for toxicities without safety risk as determined by the investigator, such as alopecia, Grade 2 peripheral neurotoxicity associated with prior platinum therapy, etc.).
9. Organ function shall meet the following requirements:

   1. No blood products, hematopoietic cell growth factors (e.g., granulocyte colony stimulating factor, erythropoietin), or other medication received to correct abnormal blood routine at least 2 weeks before initial administration, and blood routine: Absolute neutrophil count (ANC) ≥1.5×109/L, Platelets (PLT) ≥100×109/L, Platelets (Hb) ≥90g/L;
   2. Pancreatic function: Serum total amylase ≤1.5× upper limit of normal (ULN); Serum lipase ≤1.5×ULN (it is allowed to be included if serum total amylase>1.5× ULN, but the pancreatic amylase is in the ULN range);
   3. Hepatic function: Total serum bilirubin (TBIL) ≤ 1.5×ULN, Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5×ULN if no liver metastases, or otherwise TBIL ≤ 3×ULN, AST and ALT ≤ 5×ULN.
   4. Renal function: Creatinine clearance ≥ 50 mL/min (according to Cockcroft-Gault Equation).
   5. Coagulation function: International normalized ratio (INR) and prothrombin time (PT)≤ 1.5×ULN (except for patients receiving anticoagulant therapy).
10. Be able to swallow medication, follow protocol procedures, and comply with follow-up visit requirements.
11. Female patients with reproductive potential agreed to use effective method of contraception throughout the entire study duration and for at least 3 months after the last dose of study medication.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible to participate in this study:

1. Patients with known driver alterations other than ALK, such as EGFR, MET, RET, ROS1, NTRK, etc. (If ALK co-mutation exists, the patient can discuss with the investigator for enrollment);
2. Previous treated with any third-generation ALK TKI (including marketed drugs such as loratinib, and unmarketed investigational drugs);
3. History of allergy to any component or excipient of SY-3505 capsules;
4. With other primary malignancies, except those that have been cured and have not recurred within 2 years prior to screening, and those that have been cured of basal or squamous cell carcinoma of the skin, carcinoma in situ of cervix, or carcinoma in situ of breast;
5. The presence of symptomatic primary CNS tumors, symptomatic CNS metastases, leptomeningeal carcinomatosis, or untreated spinal cord compression. Except: Patient had stable CNS disease (no evidence of progression identified by imaging for at least 4 weeks prior to initial administration, and all neurological symptoms had recovered to baseline), no evidence of new or progressive brain metastases, no CNS surgery or radiotherapy within 4 weeks prior to initial administration, and no stereotactic radiosurgery (SRS) within 2 weeks prior to initial administration. Steroid administration was stopped or the dose stabilized within 2 weeks prior to initial administration. (This exception does not include cancerous meningitis, which should be excluded regardless of clinically stable conditions).
6. The following symptoms or diseases occurred prior to initial administration and remain poorly controlled after optimal treatment:

   1. Systemic bacterial, viral or fungal infection with uncontrolled activity;
   2. Poorly controlled (poorly control refers to the effusion increases significantly within 2 weeks after extraction, with obvious symptoms, requiring further puncture or other intervention) pleural effusion, abdominal effusion or pericardial effusion after intervention (such as drainage) ;
   3. Poorly controlled diabetes (fasting blood glucose ≥11.1 mmol/L and/or HbA1c ≥ 8%);
   4. Uncontrolled symptomatic hyperthyroidism or hypothyroidism as assessed by the investigator;
   5. Uncontrolled electrolyte disturbances (e.g., hypocalcemia, hypomagnesium, hypokalemia) as assessed by the investigator;
   6. Clinically significant gastrointestinal disorders included active ulcerative colitis, Crohn's disease, gastrointestinal ulcers, or prior surgical procedures that could significantly affect drug absorption as assessed by the investigator.
7. Presence with severe cardiovascular diseases/abnormalities, meeting any of the following criteria:

   1. Patients with corrected QT interval for heart rate according to Fridericia's formula > 470 msec (females) and > 450 msec (males) during the screening period (If prolonged QTcF suspected to be caused by medication and was assessed as safe and controllable by the investigator, the patient can be enrolled after drug correction);
   2. Left ventricular ejection fraction (LVEF) < 50%;
   3. Myocardial infarction or unstable angina or clinically significant uncontrolled arrhythmias, including bradyarrhythmia (such as type II second degree heart block or third degree heart block) that may lead to prolonged QTcF within 6 months prior to initial administration;
   4. Class III or IV congestive heart failure according to New York Heart Association (NYHA) classification;
   5. History of poorly controlled hypertension, unstable hypertension, or poor compliance with antihypertensive therapy as assessed by the investigator.
8. Presence or with histiory of the following active viral infection:

   1. Active hepatitis B (HBsAg positive and HBV-DNA ≥2×103 IU/mL, patients could be included if the HBV-DNA value decreased to below 2×103 IU/mL after regular antiviral therapy) or active hepatitis C virus infection (HCV-RNA >ULN on central test) at screening;
   2. HIV positive at the time of screening or have a known history of other immunodeficiency diseases;
   3. History of organ transplantation, hematopoietic stem cell or bone marrow transplantation.
9. Presence of other lung diseases that require systematic therapy or are severe, such as active tuberculosis, interstitial lung disease, etc., that may affect the interpretation of the study results or put patients at high risk according to the judgment of the investigator;
10. Have used CYP3A4 potent inhibitors (atazanavir, clarithromycin, Indinavir, Itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telomycin, troleandomycin, voriconazole, grapefruit [juice]) or inducers (carbamazepine, phenobarbital, phenytoin, rifabutin, St. John's Wort, Rifampicin) within 2 weeks prior to initial administration or cannot be stopped during the study;
11. The following antitumor treatments were administered prior to initial administration: More than 30% of bone marrow radiation or extensive radiotherapy (within 4 weeks prior to initial administration); Palliative radiotherapy (within 7 days prior to initial administration); Other antitumor agents treatment (within 2 weeks prior to initial administration or within 5 half-life times of the agent, whichever is longer), such as chemotherapy, targeted therapy (immunotherapy or other antibody-based therapies).
12. Major surgery (defined as Grade ≥3 surgery, excluding central venous catheter placement, tumor punch biopsy, and gastric tube placement) or significant trauma within 4 weeks prior to initial administration, and did not fully recover.
13. Have participated in other clinical studies within 4 weeks prior to initial administration (Note: Patients who did not use the investigational drug or investigational medical device or who had discontinued treatment from other clinical studies and only followed up for survival were excluded) or plan to participate in other clinical studies during the study.
14. History of severe arteriovenous thrombosis (such as cerebrovascular accident [including transient ischemic attack], deep vein thrombosis, and pulmonary embolism) within 1 year prior to initial administration and has the potential to increase the risk in the study as assessed by the investigators, or a tendency to bleed within 30 days prior to initial administration, or a risk of major gastrointestinal bleeding as determined by the investigators.
15. Pregnant or lactating woman.
16. Other conditions assessed unsuitable for participation in this study, such as other serious acute or chronic diseases, or laboratory abnormalities that may increase the risk for the patient, or may interfere with interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) assessed by the independent review committee (IRC) | Up to 2 years
  ORR is defined as the proportion of patients achieving an objective response (complete response [CR] or partial response [PR]) according to Response Evaluation Criteria in Solid Tumors (RECIST), v.1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
ORR assessed by the investigator | Up to 2 years
  ORR is defined as the proportion of patients achieving an objective response (CR or PR) according to RECIST 1.1.
Disease Control Rate (DCR) assessed by the investigator and IRC | Up to 2 years
  DCR is defined as the proportion of patients achieving an objective response (CR or PR) or stable disease (SD) according to RECIST 1.1.
Progression-Free Survival (PFS) assessed by the investigator and IRC | Up to 2 years
  PFS is defined as the time interval from the date of the first dose of the study treatment until the first date at which disease progression is objectively documented, or death due to any cause, whichever occurs first. PFS will be censored for participants without documented disease progression or death.
Time to Tumor Response (TTR) assessed by the investigator and IRC | Up to 2 years
  TTR is defined as the time from the first dose and the first occurrence of an objective response (CR or PR) based on RECIST 1.1.
Duration of Response (DoR) assessed by the investigator and IRC | Up to 2 years
  DoR is defined as the time from the first occurrence of an objective response (CR or PR), based on RECIST 1.1 to first documented disease progression or death.
Intracranial Objective Response Rate (IC-ORR) assessed by the investigator and IRC | Up to 2 years
  IC-ORR is defined as the proportion of patients with intracranial target lesions that are measurable at baseline who achieve an objective response (CR or PR) according to RECIST 1.1 and Revised Assessment in Neuro Oncology (RANO) criteria.
Intracranial Disease Control Rate (IC-DCR) assessed by the investigator and IRC | Up to 2 years
  IC-DCR is defined as the proportion of patients with intracranial target lesions that are measurable at baseline who achieve an objective response (CR or PR) or SD according to RECIST 1.1 and Revised Assessment in Neuro Oncology (RANO) criteria.
Intracranial Duration of Response (IC-DoR) assessed by the investigator and IRC | Up to 2 years
  IC-DoR was defined as time from documentation of intracranial response (CR or PR) to intracranial disease progression or death.
Overall Survival | Up to 2 years
  OS is defined as the time interval from the date of the first dose of the study treatment until death due to any cause. It will be censored on the date of last contact for those participants who are alive.
Incidence of Treatment-emergent adverse events (AEs) and serious adverse events (SAEs) as characterized and graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event [CTCAE] v5 | Up to 2 years
  To evaluate safety and tolerability of the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Sun, Study Director — Shouyao Holdings (Beijing) Co. LTD
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China